CLINICAL TRIAL: NCT04919109
Title: Phase 1, Randomized, Double-blind, Placebo-controlled, Dose-escalation Study Evaluating Safety and Immunogenicity of CodaVax-RSV in Seropositive and Seronegative Children
Brief Title: Safety and Immunogenicity of CodaVax-RSV in Seropositive and Seronegative Children
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Codagenix, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CDX-RSV-101P
Record Dates: First submitted 2021-05-26; First posted 2021-06-09 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: RSV; Live-attenuated vaccine; respiratory infection; Pediatric; Codon-deoptimized
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Respiratory Tract Infections | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo comparator (Placebo Comparator): Administered as nose drops
  Interventions: Biological: Normal Saline
- Experimental: CodaVax-RSV 10^6 PFU (Experimental): Respiratory syncytial virus live attenuated vaccine against RSV administered as nose drops
  Interventions: Biological: CodaVax-RSV
- Experimental: CodaVax-RSV 10^5 PFU (Experimental): Respiratory syncytial virus live attenuated vaccine against RSV administered as nose drops
  Interventions: Biological: CodaVax-RSV
- Experimental: CodaVax-RSV 10^4 PFU (Experimental): Respiratory syncytial virus live attenuated vaccine against RSV administered as nose drops
  Interventions: Biological: CodaVax-RSV
- Experimental: CodaVax-RSV 10^3 PFU (Experimental): Respiratory syncytial virus live attenuated vaccine against RSV administered as nose drops
  Interventions: Biological: CodaVax-RSV

INTERVENTIONS:
Biological: CodaVax-RSV — live attenuated vaccine against RSV
  Arms: Experimental: CodaVax-RSV 10^3 PFU; Experimental: CodaVax-RSV 10^4 PFU; Experimental: CodaVax-RSV 10^5 PFU; Experimental: CodaVax-RSV 10^6 PFU
Biological: Normal Saline — Placebo comparator
  Arms: Placebo comparator

SUMMARY:
This study is a Phase 1, randomized, double-blind, placebo-controlled, dose-escalation clinical trial to evaluate the safety of and immune response to CodaVax-RSV in healthy children. They will be vaccinated in spring to early autumn 2023 and followed through the 2023-24 RSV season. 18 children aged 2 to 5 years who are RSV-seropositive (have antibodies to RSV) and 33 children aged 6 months to < 2 years who are RSV-seronegative (do not have antibodies to RSV) will be enrolled in escalating-dose cohorts. A safety committee will review the safety profile of each dosing group before the next dose-escalation. Children will receive 2 doses of the vaccine at one of several dose levels or placebo (saline solution with no active ingredient) as nose drops; doses will be 28 days apart.

A parent/guardian will record temperature and other conditions in a diary daily for 7 days after each dose. The parent/guardian will be contacted by telephone on the day after Dose 1 for safety assessment and review of the diary data. Children will return to the clinic 3, 7, 14, and 28 days after each dose. The parent/guardian will then be contacted by telephone monthly until 1 year after the second dose.

Study procedures include physical examinations, vital signs, and collections of blood and nose/throat swab samples to look at safety of the vaccine and to analyze body's immune response.

ELIGIBILITY:
Inclusion Criteria:

1. Age at the time of informed consent:

   * Part A: 2 to 5 years, inclusive
   * Part B: 6 months to < 2 years
2. RSV Status at Screening:

   * Part A: RSV-seropositive
   * Part B: RSV-seronegative
3. Good general health status
4. Product of normal full-term pregnancy (36 to 42 weeks gestation)

Exclusion Criteria:

1. Household contact with any of the following groups of individuals for the period up to 14 days after each dose:

   * Pregnant women
   * Infants < 6 months of age
   * With hospitalization for asthma or other chronic respiratory disease in the past 5 years
   * Immunocompromised individuals, which includes, but is not limited to, those with the following conditions:

     * AIDS
     * Receipt of chemotherapy within the past 6 months
     * Current receipt of immunosuppressive agents
     * Solid organ or bone marrow transplant
2. Enrolled in the same classroom at full-time day care with infants < 6 months of age for 14 days after each dose
3. Household contact of another child enrolled into the study
4. Inadequate venous access for repeated phlebotomy
5. Height and weight ≤ 5th percentile for age and sex (according to CDC growth charts for children in Part A, according to World Health Organization Child Growth Standards for children in Part B)

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-08-27 (Estimated)

PRIMARY OUTCOMES:
Number of participants reporting expected adverse reactions | Day 7
  Reactogenicity Event Counts
Number of participants reporting expected adverse reactions | Day 36
  Reactogenicity Event Counts
Number of participant reported adverse events | Days 57
  Adverse event counts
Number of participants with Medically attended AEs (MAAEs), new-onset chronic illnesses (NCIs), and serious AEs (SAEs) | Days 210
  counts

SECONDARY OUTCOMES:
Neutralizing antibody | Screening, Days 29 and 57
  Neutralizing antibody level

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Velocity, Lincoln, Nebraska
  - Velocity, Omaha, Nebraska
  - Velocity, Providence, Rhode Island
  - Velocity, West Jordan, Utah
- University of Witwatersrand (WITS)/Vaccines and Infectious Diseases Analytics (VIDA), Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: No